CLINICAL TRIAL: NCT01463449
Title: "Influence of Obesity, Weight Loss, and Diet on Low Grade Inflammation With Particular Focus on the Macrophage Marker, Soluble-CD163 - a New Predictor of Diabetes.Can s-CD163 Discriminate Between Healthy and Unhealthy Obese Individuals?"
Brief Title: "Can Soluble-CD163 Discriminate Between Healthy and Unhealthy Obese Individuals?"
Acronym: sCD163
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Novo Nordisk A/S (Industry); The Danish Medical Research Council (Other)
Responsible Party: Sponsor
Other Study IDs: 17913
Record Dates: First submitted 2011-10-26; First posted 2011-11-01 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Obesity; Insulin Resistance; Type 2-diabetes; Inflammation
Keywords: Obesity; Soluble-CD163; Macrophage; Inflammation
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus, Type 2; Inflammation | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, adipose tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Obese: Obese subjects half with type 2-diabetes. Before and after gastric bypass. Expected reduction in weight 25 %. We expect a reduction in low grade inflammation in adipose tissue after weight loss.
  Interventions: Procedure: gastric bypass

INTERVENTIONS:
Procedure: gastric bypass — Low grade inflammation in adipose tissue before and after gastric bypass
  Other Names: Soluble-CD163

SUMMARY:
CD163 is a membrane bound receptor primary expressed in monocytes and macrophages. A soluble variant of CD163 (sCD163) is present in plasma and is elevated in pathological condition activating the monocyte-macrophage system. Recently sCD163 is associated with various inflammatory conditions, ex. adipose tissue inflammation and very recently to be a rather strong predictor of the development of type 2-diabetes. Only a subset of obese individuals develops insulin resistance, type 2-diabetes and related diseases. These healthy obese subjects are characterized of less adipose tissue inflammation and less insulin resistance as compared to unhealthy obese individuals. Consequently it would be of great importance to develop markers that could discriminate between healthy and unhealthy obese subjects. Aim: To investigate whether macrophage CD163 is involved in adipose tissue inflammation in obesity and thereby to the metabolic complications of metabolic syndrome. To investigate how sCD163 is regulated by metabolic factors such as obesity, fat distribution, weight loss and diet. Methods: Intervention study. 45 morbidly obese subject approved to gastric by-pass. Blood samples, MR-spectroscopy, DXA, weight control and fat biopsy are taken before and 12 month after surgery. Correlations studies: to investigate the influence of diet and weight loss on CD163 and sCD163. Perspective: To study the role of macrophages infiltration and activation for adipose tissue inflammation and to determine whether the macrophage marker, s-CD163, together with other markers will be able better to identify obese individuals who are at increased risk for developing complications such as diabetes

DETAILED DESCRIPTION:
It is recognized that low grade inflammation is a key player in the development of atherosclerosis and insulin resistance (Haslam, James 2005). Circulating levels of inflammatory markers such as high sensitive C-reactive protein (hsCRP) and interleukin (IL)-6 are found to be increased in subjects with cardiovascular disease (CVD) and type 2-diabetes (Dandona, Aljada & Bandyopadhyay 2004). We and others have shown that obesity, and in particular abdominal obesity, is associated with persistent increased level of inflammatory markers (Bruun et al. 2007, Christiansen et al. 2010a) . Thus this low grade of inflammation may represent "the common soil" for the pathogenesis of atherosclerosis and insulin resistance and represent the link between these metabolic disturbances and obesity.

Besides its function as a storage organ, the adipose tissue (AT) exerts a complex role in the organism. In obesity the adipose tissue is infiltrated by an increased amount of macrophages, and particular these macrophages express and release a wide range of hormones and cytokines, collectively called adipokines, which biological functions are shown to include involvement in glucose metabolism, lipid metabolism, adipocyte differentiation, immunity, vasculature and neuron development and eating behavior (Trayhurn, Wood 2004).

Among the adipokines expressed in the AT are pro-inflammatory cytokines as TNFα, IL-6, pro-inflammatory chemokines as IL-8, MCP-1, MIP1α, thrombotic factors as plasminogen inhibitor 1 (PAI-1), and AT specific proteins as adiponectin and leptin.

Hypertrophied adipocytes, as seen in obese subjects and associated with insulin resistance are shown to display a distinct gene expression of inflammatory markers compared to small human adipocytes and it is shown that adipocyte size is an important determinant of adipokine secretion. Moreover an positive association between the grade of obesity and the expression of pro-inflammatory cytokines as TNFα, IL-6, IL-8, has been found whereas and an inverse association between adiponectin and obesity has been reported (Kern et al. 2003, Bruun et al. 2003).In accordance with these observations, we have found the AT expression of MCP-1 was up-regulated in obese subjects (Christiansen, Richelsen & Bruun 2005) whereas the AT expression of adiponectin in obese subjects (mean BMI 40 kg/m2 ) was found down-regulated with 50% as compared to lean subjects (mean BMI 22 kg/m2) (Christiansen et al. 2010b).

Thus, adipose tissue inflammation resulting in dysfunction of the adipose tissue may be the important factor relating obesity to insulin resistance, metabolic syndrome, diabetes, and cardiovascular diseases.

CD163:

CD-163 is a membrane bound receptor primary expressed in monocytes and macrophages. CD163 was originally described as a hemoglobin scavenger receptor since it is involved in removing hemoglobin released from ruptured red blood cells (Moestrup, Moller 2004). A soluble variant of CD-163 (s-CD-163) is present in plasma and is elevated in pathological condition activating the monocyte-macrophage system.

Recently s-CD-163 is associated with various inflammatory conditions (Moestrup, Moller 2004), and very recently to be a rather strong predictor of the development of type 2 diabetes in a large Danish cohort (Moller et al. 2011). Thus, s-CD-163 may be a marker both related to inflammation as well as to metabolic conditions maybe linking low grade inflammation and metabolic abnormalities, and furthermore, may be a marker of the obese state with complications.

Only a subset of overweight and obese individuals develops insulin resistance, type 2 diabetes and related diseases (Stefan et al. 2008, Bluher 2010). These "healthy" obese subjects are characterized of less adipose tissue inflammation and less insulin resistance as compared to unhealthy obese individuals. Consequently it would be of great importance to develop markers or predictors that could discriminate between "healthy" and unhealthy obese subjects in order to made a better selection for more invasive treatment such as e.g. surgery, pharmacotherapy etc.

Research Plan:

1. Is CD163 pathophysiologically involved in adipose tissue inflammation in obesity? Adipose tissue (AT) is taken from various regions in lean to very obese subjects - from either subcutaneous fat biopsies (lean subjects), surgery (obese subjects - BMI> 30), and from bariatric surgery (gastric bypass) in the very obese subjects (BMI > 40) - both subcutaneous and visceral AT are investigated in parallel in the very obese individuals.

   In the adipose tissue the amount of macrophages will be determined by both biochemical (e.g. CD68) and microscopically methods (immunohistochemistry). Moreover, the gene expression (PCR) and protein (Western blot) of CD163 will be detected in AT and related to the expression and protein of a number of other proinflammatory adipokines.
2. Is s-CD163 a marker of adipose tissue inflammation and metabolic disturbances? Blood samples from the individuals in project 1 will also be obtained and s-CD163 measured (in house sandwich ELISA kit (Moller, Hald & Moestrup 2002)). These values will be related to the amount of macrophages in AT and the expression of CD136 in AT. Moreover, the insulin sensitivity determined by the HOMA model will be performed, and s-CD163 related to the HOMA score.
3. Is s-CD163 affected by weight loss, and dietary changes ( e.g. the effect of fructose (proinflammatory) and the effect of resveratrol (antiinflammatory)?

   1. Weight loss will be induced by bariatric surgery (bypass) in very obese subjects (BMI > 40). S-CD163 and changes in insulin sensitivity (HOMA) and other inflammatory markers (e.g. hsCRP, IL-6, TNF, MCP-1, adiponectin etc.) will be measured before and after 6 and 12 months after surgery. From power calculations it is planned to include 45 very obese subjects in this study - half of them with type 2 diabetes.
   2. We have performed dietary investigations with fructose (soft drinks taken for 6 months in 50 overweight and obese subjects) which induces ectopic fat accumulation in the liver determined by MR-spectroscopy and insulin resistance, and dietary intervention with resveratrol which reduces liver fat and has antiinflammatory effects. In frozen plasma samples from these studies s-CD163 will be measured in order to get insight in the dietary effect of fructose and resveratrol on this and related markers.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* Legally competent (Habil)
* Age 30-60
* Approved to gastric bypass, according to current criteria in Denmark
* Written consent
* Investigators verification of the suitability

Exclusion Criteria:

* Heart, liver or kidney disease
* Treatment with cortisol
* MR-contraindications
* Abuse/addiction
* Malignancy
* Weight more than 145 kg because of problems with DXA and MRI

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The cohorts will be selected from the department of Endokrinology at Aarhus University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Low grade inflammation in adipose tissue after weight loss induced by gastric bypass | Primary endpoint after 12 months.
  sCD163 measured by enzyme-linked immunosorbent assay (ELISA). And CD163 gene expression measured by Real Time PCR (RT-PCR).

SECONDARY OUTCOMES:
Quantity of fat in the liver | 12 months.
  The quantity of fat in the liver at baseline and again 12 months after surgery. Assessed by MR spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Richelsen, Prof. Dr.Med, Study Director — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Endocrinology, Aarhus University Hospital, Aarhus
  - Department of Endocrinology, Aarhus University Hospital, Aarhus C